CLINICAL TRIAL: NCT05148507
Title: Optimization of the Ocular Surface Prior to Cataract Surgery Using PROKERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Wongskhaluang (Other)
Responsible Party: Sponsor-Investigator, Jeff Wongskhaluang, Physician, Principal Investigator, Grin Eye Care
Organization: Grin Eye Care (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9132
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cataract; Dry Eye Syndromes; Cataract Senile; Dry Eye
MeSH Terms: conditions — Cataract; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Application of cryopreserved amniotic membrane (Prokera)
  Interventions: Device: PROKERA

INTERVENTIONS:
Device: PROKERA — Amniotic membrane is the sac that encloses the baby during pregnancy. Amniotic membrane has been used to treat many ocular (eye) diseases and repair ocular surface damage. PROKERA contains amniotic membrane fastened between a ring system and can be worn in the eye like a contact lens. PROKERA is a medical device that was cleared by the United States food and drug administration (FDA) in 2003.

SUMMARY:
The purpose of the study is to assess whether PROKERA can sufficiently stabilize the ocular surface prior to cataract surgery and improve post operative outcomes patients with moderate to severe dry disease.

DETAILED DESCRIPTION:
Amniotic membrane has been used to treat many ocular diseases and repair ocular surface damage. PROKERA contains amniotic membrane fastened between a ring system and can be worn in the eye like a contact lens. PROKERA is a medical device that was cleared by the United States Food and Drug Administration (FDA) in 2003.

Cataract surgery is the most common eye surgery done in the United States. Prior to cataract surgery, machines scan the eyes to calculate which implant is needed at the time of cataract surgery. When a patient has dry eyes, the machines may have inaccurate measurements.

The purpose of the study is to assess whether PROKERA can sufficiently stabilize the ocular surface prior to cataract surgery and improve post operative outcomes patients with moderate to severe dry disease. There will be a maximum of 64 eyes of individuals age 18 and older in the study enrolled at one study site. Each subject will have both eyes evaluated for the study.

Prior to cataract surgery, patients enrolled in the study will have PROKERA device inserted on the surface of the eye. The subject will then come back after about five days to remove the PROKERA device and follow up again in one week and two weeks after the removal of the PROKERA device. During both of the follow up visits, the study doctor will grade symptoms based on a questionnaire, examine eyes, take pictures, and grade the severity of the dry eye disease to determine any changes from the baseline testing.

At the two week visit, cataract surgery will be scheduled, which will be within one to two weeks time. After surgery, a one month postoperative visit will occur, where the same examination procedures are performed as the previous follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age and plan to undergo cataract surgery
2. Prior use of DED/keratitis conservative treatments (artificial tears, ointment, Xiidra®, Restasis, warm compresses, etc.) within 30 days
3. Moderate to severe DED/keratitis (SPEED score ≥ 10)
4. Total cornea fluorescein staining score ≥ 4 (NEI scale)
5. Topographic changes such as irregularity, dropout, and higher order aberrations (HOAs; RMS > 0.4) as determined by the investigator
6. Distorted keratometry mires or inconsistent biometry between 2 consecutive readings (30s apart) as determined by the investigator

   Exclusion Criteria:
7. Use of soft contacts lens, bandage contact lens, or scleral lens within 7 days
8. Ocular surgery within 3 months
9. History of refractive surgery (LASIK, keratectomy, radial keratotomy, etc.)
10. History of clinically significant ocular trauma
11. Significant posterior corneal astigmatism (≥ 0.75 D)
12. History of herpetic keratitis
13. Ongoing ocular or systemic infection
14. Visually significant retinal pathology
15. Clinically significant findings observed at screening, including lid abnormalities, epithelial basement membrane dystrophy, Salzmann's nodular degeneration, subclinical or clinical keratoconus (defined as KISA% index > 6019), ectasia (Belin/Ambrosio enhanced ectasia display final 'D' index > 2.6920), Fuchs' endothelial corneal dystrophy (Using the Classification by Sun et al21), etc.
16. Short eyes (axial length < 22 mm22, 23)
17. High myopia (axial length ≥ 26 mm)22, 24
18. Eyes with glaucoma drainage devices or filtering bleb
19. Patients with a history of drug reactions to Ciprofloxacin, Amphotericin B, Glycerol, and/or DMEM.
20. Patient cannot close the eyelid, has an incomplete blink, or demonstrates any other signs of exposure that cannot be addressed by the investigator
21. Pregnancy or subject expecting to be pregnant
22. Use of additional eye medications (i.e. glaucoma eye drops, anti-histamines, etc)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Percentage to achieve emmetropia | 2-3 months
  Defined as spherical equivalent -0.5D to +0.5D and <1.0D astigmatism before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Grin Eye Care, Olathe, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided